CLINICAL TRIAL: NCT04752111
Title: Dose Esmolol Infusion Have an Adjuvant Effect to Transversus Abdominis Plane Block for Pain Control in Laparoscopic Cholecystectomy: A Randomized Controlled Double-blind Trial.
Brief Title: Dose Esmolol Infusion Have an Adjuvant Effect to TAP Block for Pain Control in Laparoscopic Cholecystectomy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Samar Rafik Mohamed Amin, lecturer of anesthesia and surgical ICU, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC3-12-2020
Record Dates: First submitted 2021-01-28; First posted 2021-02-12 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain
Keywords: Esmolol infusion; TAP block; cholecystectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — esmolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group E (esmolol infusion) (Experimental): 10 minutes before induction of anesthesia the patients will receive a loading dose of injection esmolol 0.5 mg/kg in 30 ml isotonic saline in the IV line, followed by an IV infusion of esmolol 0.05 mg/kg/min till the completion of surgery After induction of anesthesia and before starting the surgery, patients will receive bilateral in-plane ultrasound guided transversus abdominis plane block with 40 ml of bupivacaine 0. 25% after induction of anesthesia 20 ml in each side .
  Interventions: Drug: Esmolol
- Group T (TAP block) (Placebo Comparator): 10 minutes before induction of anesthesia the patients will receive a loading dose of injection 30 ml isotonic saline in the iv line, followed by an IV infusion of saline at a rate of 0.05 mg/kg/min till the completion of surgery After induction of anesthesia and before starting the surgery, patients will receive bilateral in-plane ultrasound guided transversus abdominis plane block with 40 ml of bupivacaine 0. 25% after induction of anesthesia 20 ml in each side.
  Interventions: Drug: Esmolol

INTERVENTIONS:
Drug: Esmolol — administration of a loading dose esmolol infusion 0.5 mg/kg in 30 ml isotonic saline in the IV line, followed by an IV infusion of esmolol 0.05 mg/kg/min till the completion of surgery

SUMMARY:
Pain after laparoscopy differs considerably from that seen after laparotomy. Laparotomy results mainly in parietal pain (abdominal wall), where as Pain in laparoscopy results from stretching of the intra-abdominal cavity, peritoneal inflammation, and diaphragmatic irritation caused by residual carbon-dioxide in the peritoneal cavity. The transverse abdominis plane (TAP) block is a peripheral nerve block designed to anesthetize the nerves supplying the anterior abdominal wall (T6 to L1). While esmolol is an ultra-short acting intravenous β-blocker having a rapid onset and offset effect. It provides an unprecedented level of tolerability and safety in the perioperative setting. When used as an adjunct, it has been shown to improve the postoperative recovery by reducing postoperative pain intensity and intraoperative anesthetic and opioid requirements and preventing opioid-induced hyperalgesia . The mechanism of this synergistic effect is uncertain, but both pharmacokinetic and pharmacodynamics interactions with anesthetic drugs have been proposed.

ELIGIBILITY:
Inclusion Criteria:

1. ASA grade I/II patients undergoing laparoscopic cholecystectomy .
2. Age group of 18 -60 years.
3. Patients giving valid informed consent.

Exclusion Criteria:

1. Patient refusal
2. Patients belonging to ASA grade III and grade IV .
3. Coagulation disorders.
4. Patients with known allergy to one of the used drugs.
5. Extreme obesity (BMI >35)
6. Patients with cardiac, pulmonary, hepatic or renal disorders
7. Pregnancy
8. Drug abusers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
pain rescue-analgesia consumption | 24 hours postoperative
  . If pain score exceed 3, rescue analgesia 5 mg bolus of morphine will be administered intravenous to achieve satisfactory pain control that can be repeated every 4-6 hours.

SECONDARY OUTCOMES:
Visual analogue pain score | every 0,2,4,6,12, up to 24 hours postoperative
  scales from zero (no pain) to ten (unbearable pain)
Intraoperative hemodynamic data | 30 minutes after induction of anesthesia
  mean arterial blood pressure and heart rate
Postoperative nausea and vomiting | 24 hours postoperative
  A three-point rating scale (1: no postoperative nausea and vomiting, 2: nausea without vomiting, 3: nausea with vomiting. Ondansetron 4 mg will be available if required.
Patient satisfaction | 24 hours postoperative
  using a 5-point Likert scale (1 was "very unsatisfied", 2- "unsatisfied", 3- "unsure", 4- "satisfied", and 5- "very satisfied").

CONTACTS AND LOCATIONS:
Locations (1):
- Samar Rafik Mohamed Amin, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided